CLINICAL TRIAL: NCT01376518
Title: Influence of Positive End-expiratory Pressure on the Cerebrovascular Autoregulation in Patients With Respiratory Failure
Brief Title: Influence Positive End-expiratory Pressure on Autoregulation in Patients With Respiratory Insufficiency
Acronym: dARICUPEEP
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Patrick Schramm, Senior Physician, Johannes Gutenberg University Mainz
Other Study IDs: 837.041.10 1
Record Dates: First submitted 2011-06-14; First posted 2011-06-20 (Estimated); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Respiratory Insufficiency
Keywords: acute respiratory distress syndrome; acute lung injury; cerebrovascular autoregulation; transcranial Doppler; ventilation
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Distress Syndrome; Acute Lung Injury; Respiratory Aspiration | interventions — Positive-Pressure Respiration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- respiratory failure: patients with respiratory failure and need of high positive end-expiratory pressure ventilation.
  Interventions: Procedure: positive end-expiratory pressure

INTERVENTIONS:
Procedure: positive end-expiratory pressure — Elevation of positive end-expiratory failure for recruitment
  Other Names: PEEP

SUMMARY:
The aim of the present study is to characterize the influence of an elevated positive end-expiratory pressure in patients with acute respiratory distress syndrome or acute lung injury on the cerebrovascular autoregulation.

DETAILED DESCRIPTION:
Cerebral blood flow velocity will be measured using transcranial Doppler sonography and then correlate with the invasive arterial blood pressure curve to calculate the index of cerebrovascular autoregulation Mx (Mx>0.3 indicates impaired AR). The index of cerebrovascular autoregulation Mx was measured during baseline positive end-expiratory pressure (PEEP) levels and after lung recruitment with higher level of PEEP. The equality between this two PEEP levels was estimated and calculated with one side Wilcoxon test.

ELIGIBILITY:
Inclusion Criteria:

* respiratory failure
* Age >18 years
* Invasive ventilation

Exclusion Criteria:

* Sepsis
* preexisting cerebral illness
* traumatic brain injury
* meningitis or encephalitis
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients on intensive care unit with acute respiratory failure
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Integrity of the cerebrovascular autoregulation (CA) | 30 Minutes
  Cerebrovascular autoregulation will be calculated as a moving correlation index (Mx) from the cerebral blood flow velocity and the arterial blood pressure. It is a parameter without unit (index).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Schramm, MD, Principal Investigator — Department of Anesthesiology, University medicine Mainz, Germany
Locations (1):
- University medical centre, Mainz, Germany

REFERENCES:
- [Result] Schramm P, Closhen D, Felkel M, Berres M, Klein KU, David M, Werner C, Engelhard K. Influence of PEEP on cerebral blood flow and cerebrovascular autoregulation in patients with acute respiratory distress syndrome. J Neurosurg Anesthesiol. 2013 Apr;25(2):162-7. doi: 10.1097/ANA.0b013e31827c2f46. PMID 23211642